CLINICAL TRIAL: NCT07385833
Title: Disaster Preparedness in Patients With Diabetic Foot: The Effect of an Educational Intervention
Acronym: Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Senem Duman (Other)
Responsible Party: Sponsor-Investigator, Senem Duman, Lecturer, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SaglikBilimleriU-3
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Foot; Type 2 Diabetes Mellitus
Keywords: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disaster Preparedness Education Program (Other): The intervention consists of two face-to-face theoretical education sessions delivered over two weeks. Week 1 includes a 2-hour session on diabetic foot management (definition, risk factors, care principles) supported by visual materials and interactive Q&A. Week 2 includes a session on disaster and emergency management for individuals with diabetic foot, covering preparedness before disasters, actions during disasters, and post-disaster strategies to protect foot health. The contents of an emergency kit/go-bag are physically demonstrated, and participants are asked to prepare their own kit and bring it to the next visit. At post-test, emergency kits/go-bags are inspected using a standardized checklist and feedback is provided for missing or incorrect items.
  Interventions: Behavioral: Disaster Preparedness Education Program
- Routine Care (Control) (No Intervention): Participants receive routine diabetes care and follow-up as provided by the institution. No structured education on disaster preparedness or foot self-care behaviors is delivered during the study period. Data are collected at the same time points as the intervention group.

INTERVENTIONS:
Behavioral: Disaster Preparedness Education Program — The intervention consists of two face-to-face theoretical education sessions delivered over two weeks. Week 1 includes a 2-hour session on diabetic foot management (definition, risk factors, care principles) supported by visual materials and interactive Q&A. Week 2 includes a session on disaster and emergency management for individuals with diabetic foot, covering preparedness before disasters, actions during disasters, and post-disaster strategies to protect foot health. The contents of an emergency kit/go-bag are physically demonstrated, and participants are asked to prepare their own kit and bring it to the next visit. At post-test, emergency kits/go-bags are inspected using a standardized checklist and feedback is provided for missing or incorrect items.
  Arms: Disaster Preparedness Education Program

SUMMARY:
This quasi-experimental study aims to evaluate the effect of a disaster preparedness education program on disaster preparedness levels, foot care behaviors, and diabetic foot care self-efficacy in patients with type 2 diabetes diagnosed with diabetic foot. Participants are assigned to an intervention group receiving structured education on diabetic foot management and disaster preparedness, or to a control group receiving routine care. Outcomes are assessed at baseline, post-intervention, and follow-up.

DETAILED DESCRIPTION:
Patients with diabetic foot are considered a vulnerable population during disasters due to disrupted access to healthcare, medications, and self-care resources. This study evaluates a structured disaster preparedness education program designed specifically for patients with diabetic foot. The intervention includes education on diabetic foot management, disaster preparedness strategies, and preparation of emergency kits and go-bags. The effects of the program on disaster preparedness, foot self-care behaviors, and self-efficacy are assessed using validated measurement tools across three time points. The findings aim to contribute to the development of disaster-focused educational interventions for individuals with chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with type 2 diabetes mellitus for at least 6 months

  * Diagnosed with diabetic foot classified as Wagner grade 1, 2, or 3
  * Receiving outpatient or inpatient care at the diabetic foot center
  * Able to communicate and complete self-report questionnaires
  * Willing to participate and provide written informed consent

Exclusion Criteria:

* • History of diabetic foot-related amputation

  * Presence of active Charcot neuroarthropathy
  * Severe cognitive impairment affecting participation
  * Significant communication barriers preventing completion of assessments
  * Presence of acute medical conditions requiring immediate intensive treatment during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Disaster Preparedness Level | Baseline, Week 3 (post-intervention), and Week 7 (follow-up)
  Disaster preparedness level is measured using the Disaster Preparedness Scale (DPS), a 15-item validated self-report scale assessing disaster physical protection, disaster planning, disaster assistance, and disaster warning and signals. Total scores range from 15 to 60, with higher scores indicating greater disaster preparedness. The primary outcome is the change in DPS total score from baseline.

SECONDARY OUTCOMES:
Change in Diabetic Foot Care Self-Efficacy | Baseline, Week 3 (post-intervention), and Week 7 (follow-up
  Diabetic foot care self-efficacy is measured using the Diabetic Foot Care Self-Efficacy Scale (DFCSES), a validated self-report scale assessing confidence in performing diabetic foot care activities. Total scores range from 0 to 100, with higher scores indicating greater self-efficacy. The outcome is the change in DFCSES total score from baseline.
Change in Foot Self-Care Behaviors | Baseline, Week 3 (post-intervention), and Week 7 (follow-up)
  Foot self-care behaviors are measured using the Foot Self-Care Behavior Scale (FSCBS), a validated 15-item scale assessing the frequency of diabetic foot care behaviors. Total scores range from 15 to 75, with higher scores indicating more positive foot self-care behaviors. The outcome is the change in FSCBS total score from baseline.
Preparation of an Emergency Kit/Go-Bag | Week 3 (post-intervention)
  Preparation of an emergency kit/go-bag is assessed by direct inspection using a standardized checklist developed according to national and international disaster preparedness guidelines. The outcome is defined as the proportion of participants who prepared a complete emergency kit/go-bag following the educational intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data are available from the corresponding author upon reasonable request

REFERENCES:
- [Result] Abbas, Z. G., & Gangji, R. R. (2025). The diabetic foot: Progress in Sub-Saharan Africa. Diabetes Research and Clinical Practice, 225, 112264. https://doi.org/10.1016/j.diabres.2025.112264 Allweiss, P. (2019). Diabetes and disasters: Recent studies and resources for preparedness. Current Diabetes Reports, 19(11), 131. https://doi.org/10.1007/s11892-019-1258-7 Alsararatee, H. H., Langley, J. C. S., Thorburn, M., Burton-Gow, H., Whitby, S., & Powell, S. (2025). Assessment of the diabetic foot in inpatients. British Journal of Nursing, 34(4), S12-S23. https://doi.org/10.12968/bjon.2024.0342 Armstrong, D. G., Tan, T. W., Boulton, A. J. M., & Bus, S. A. (2023). Diabetic foot ulcers: A review. JAMA, 330(1), 62-75. https://doi.org/10.1001/jama.2023.10578 Aziz, A. R. A., & Alsabek, M. B. (2020). Diabetic foot and disaster: Risk factors for amputation during the Syrian crisis. Journal of Diabetes and Its Complications, 34(2), 107493. https://doi.org/10.1016/j.jdiacomp.2019.107493 Bahador, R. S., Afrazandeh, S. S., Ghanbarzehi, N., & Ebrahimi, M. (2017). The impact of a three-month training programme on foot care and self-efficacy of patients with diabetic foot ulcers. Journal of Clinical and Diagnostic Research, 11(7), IC01-IC04. Bandura, A. (1977). Self-efficacy: Toward a unifying theory of behavioral change. Psychological Review, 84(2), 191-215.